CLINICAL TRIAL: NCT06298331
Title: Investigation of the Additional Effects of Aerobic Exercise Training to Abdominal Massage in Functional Constipation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SERAP ÖZGÜL, Prof. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-23073
Record Dates: First submitted 2023-11-07; First posted 2024-03-07 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Constipation
Keywords: Functional Constipation; Chronic Constipation; Abdominal Massage; Self- abdominal Massage; Aerobic Exercise; Walking; Conservative Treatment; Lifestyle Recommendation; Patient Education
MeSH Terms: conditions — Constipation | interventions — Exercise; Patient Education as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise and Abdominal Massage (Experimental): Aerobic Exercise: Aerobic exercise training will be given for 8 weeks, 3 days a week on the treadmill in the clinic under the supervision of a physiotherapist, and 8 weeks, the other 2 days a week outside the clinic. The duration of the walking session is 50 minutes (5 minutes warm-up - 40 minutes load - 5 minutes cool down).
  Abdominal Massage: Abdominal massage will be performed manually by applying baby oil to the patient's abdomen and while the patient is in the supine position. This application will take approximately 15 minutes. The massage will be performed by the physiotherapist in the clinic 3 days a week for 8 weeks and by the patient outside the clinic 2 days a week for 8 weeks as self-massage.
  Interventions: Other: Aerobic Exercise; Other: Abdominal Massage; Other: Patient Education
- Abdominal Massage (Active Comparator): Abdominal Massage: Abdominal massage will be performed manually by applying baby oil to the patient's abdomen and while the patient is in the supine position. This application will take approximately 15 minutes. The massage will be performed by the physiotherapist in the clinic 3 days a week for 8 weeks and by the patient outside the clinic 2 days a week for 8 weeks as self-massage.
  Interventions: Other: Abdominal Massage; Other: Patient Education

INTERVENTIONS:
Other: Aerobic Exercise — Aerobic exercise training will be given for 8 weeks, 3 days a week on the treadmill in the clinic under the supervision of a physiotherapist, and 8 weeks, the other 2 days a week outside the clinic. The duration of the walking session is 50 minutes (5 minutes warm-up - 40 minutes load - 5 minutes cool down). Walking speed in the clinic will be determined according to the Heart Rate Reserve(HRR) method. In the warm-up and cool-down phases in the clinic, the walking speed will be adjusted in the range of 20-40% of HRR, while in the loading phase it will be adjusted in the range of 40-60% of HRR. Heart rate will be monitored with a monitor that detects heart rate by hand contact on the treadmill. Outside the clinic, walking speed will be determined according to the level of fatigue perceived on the Borg Scale. Outside the clinic, walking speed will be regulated as 10-12 (light) on the Borg scale during warm-up and cool-down phases and 12-14 (slightly difficult) during the loading period.
  Arms: Aerobic Exercise and Abdominal Massage
Other: Abdominal Massage — Abdominal massage will be performed manually by applying baby oil to the patient's abdomen and while the patient is in the supine position. This application will take approximately 15 minutes. The massage will be performed by the physiotherapist in the clinic 3 days a week for 8 weeks and by the patient outside the clinic 2 days a week for 8 weeks as self-massage.
Other: Patient Education — Patient education will include information on the definition of constipation, causes of constipation, how constipation occurs, factors affecting constipation, concepts related to constipation, treatment options for constipation, and lifestyle recommendations for constipation, including increasing fluid intake, regulating nutrition, increasing physical activity, and regulating toilet habits.

SUMMARY:
The aim of this study was to investigate the additional effects of aerobic exercise to abdominal massage in patients with functional constipation. There are several studies investigating the effects of massage and aerobic exercise separately in functional constipation. However, to the best of our knowledge, there are no studies combining abdominal massage and aerobic exercise to demonstrate additional effects. By combining these two approaches, we believe that a higher and broader effect (local and systemic) and perhaps a cure for constipation (reaching the ideal defecation frequency or asymptomatic status) can be achieved. Therefore, this study will include individuals between the ages of 18-65 who have a diagnosis of functional constipation and who agree to participate in the study. This study is designed as a randomized controlled trial.

DETAILED DESCRIPTION:
The aim of this study was to investigate the additional effects of aerobic exercise to abdominal massage in patients with functional constipation. There are several studies investigating the effects of massage and aerobic exercise separately in functional constipation. However, to the best of our knowledge, there are no studies combining abdominal massage and aerobic exercise to demonstrate additional effects. By combining these two approaches, we believe that a higher and broader effect (local and systemic) and perhaps a cure for constipation (reaching the ideal defecation frequency or asymptomatic status) can be achieved. Therefore, this study will include individuals between the ages of 18-65 who have a diagnosis of functional constipation and who agree to participate in the study. This study is designed as a randomized controlled trial. A total of 44 individuals will be randomly assigned to 2 groups. Patients in group 1 will receive patient education with abdominal massage and aerobic exercise training. Patients in Group 2 will receive only abdominal massage and patient education. Abdominal massage and aerobic exercise will be practiced 8 weeks, 3 days a week in the clinic under the supervision of a physiotherapist, and 8 weeks, 2 days a week outside the clinic. Patient education includes information about constipation and lifestyle recommendations for constipation. Physical, sociodemographic, medical and lifestyle characteristics of the individuals will be recorded as descriptive measurements. Among the descriptive characteristics, physical activity level will be assessed with the International Physical Activity Questionnaire-Short Form and the presence of diastasis recti abdominis will be assessed with the finger width test. Outcome measures of weekly defecation frequency, defecation time, laxative use frequency and average stool consistency score will be recorded by the 7-Day Bowel Diary. Stool consistency will be questioned with the Bristol Stool Scale. Other outcome measures will be severity of constipation by the Constipation Severity Scale and Constipation Scoring System, gastrointestinal symptom level by the Gastrointestinal Symptom Rating Scale, constipation-related quality of life by the Constipation Quality of Life Scale, abdominal muscle strength by the observational/manual muscle strength test, and functional exercise capacity by the 6-min walking test. All outcome measurements will be performed at baseline and at the end of the 8th week. Perception change will be assessed using the Patient Perception of Global Change Scale, and compliance with lifestyle recommendations will be assessed using the Numeric Rating Scale. The compliance of patients with exercise and massage sessions will be assessed using diaries.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Diagnosed with chronic constipation according to Rome IV criteria
* No new treatment for constipation in the last 3 months
* Absence of any condition that would prevent compliance with the interventions and assessments in the study

Exclusion Criteria:

* Presence of secondary constipation ( uncontrolled metabolic disease (uncontrolled DM, hypothyroidism), hyperparathyroidism, neurologic disease or use of anticoagulants, anticholinergics, antihistamines, antipsychotics or opioids)
* In individuals over 50 years of age, the presence of alarm symptoms (new-onset constipation, rectal bleeding, involuntary weight loss, nausea and vomiting, fever and anemia)
* having BMI > 30 kg/m²
* having cancer diagnosis
* being pregnant or breastfeeding, being within the first year postnatally
* having irritable Bowel Syndrome, Hirschprung's Disease, Crohn's Disease, Inflammatory Bowel Disease, Megacolon diagnosis, Megarectum diagnosis, Rectocele and enterocele stage 3 and above
* presence of advanced systemic disease (e.g. cardiovascular, respiratory, renal or hepatic diseases)
* history of abdomino-pelvic or gastrointestinal surgery in the last 6 months
* presence of open wound, disruption of skin integrity, local tumor, cholestomy or abdominal hernia at the massage site
* Presence of orthopedic (e.g. lumbopelvic pain, advanced knee joint degeneration) and cardiovascular diseases (e.g. acute coronary syndrome, stage 3-4 heart valve diseases) that may prevent aerobic exercise training

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Weekly defecation frequency | Change in weekly defecation frequency from 1 week before the interventions to the end of the 1st week after the interventions.
  The bowel diary developed by Pamuk et al. is a widely used and practical diary that records defecation frequency, defecation duration, stool consistency, gas/fecal incontinence, pain during defecation and amount of laxative use. The 7-day bowel diary will be used to record weekly defecation frequency for a period of 1 week before the interventions and within 1 week following the end of the interventions

SECONDARY OUTCOMES:
Average weekly defecation time | Change in weekly duration of defecation from 1 week before the interventions to end of the 1st week after the interventions.
  The bowel diary developed by Pamuk et al. is a widely used and practical diary that records defecation frequency, defecation duration, stool consistency, gas/fecal incontinence, pain during defecation and amount of laxative use. The 7-day bowel diary will be used to record weekly defecation time for 1 week prior to the interventions and 1 week following the end of the interventions.
Average weekly frequency of laxative use | Change in weekly frequency of laxative use from 1 week before the interventions to end of the 1st week after the interventions.
  The bowel diary developed by Pamuk et al. is a widely used and practical diary that records defecation frequency, defecation duration, stool consistency, gas/fecal incontinence, pain during defecation and amount of laxative use. The 7-day bowel diary will be used to record weekly frequency of laxative use for 1 week prior to the interventions and 1 week following the end of the interventions.
Average weekly stool consistency score | Change in weekly stool consistency score from 1 week before the interventions to end of the 1st week after the interventions.
  The bowel diary developed by Pamuk et al. is a widely used and practical diary that records defecation frequency, defecation duration, stool consistency, gas/fecal incontinence, pain during defecation and amount of laxative use. In this diary, stool consistency will be questioned according to the Bristol Stool Scale. The Bristol Stool Scale, which measures colon transit time easily and quickly, was developed by Lewis and Heaton and classifies stool into 7 groups (from 1 to 7); type 1=separate hard lumps, like nuts; 2=sausage shaped but lumpy; 3=like a sausage or snake, but with cracks on its surface; 4=like a sausage or snake, smooth and soft; 5=soft blobs with clear cut edges; 6=pieces with ragged edges, a mushy stool; 7=water, no solid pieces. While type 1 and 2 indicate hard stool, type 3,4 and 5 show looser (ideal) stool. The average weekly stool consistency score will be calculated as total weekly stool consistency score / weekly frequency of defecation.
The severity of constipation and associated discomfort | Change in severity of constipation and associated discomfort from baseline up to end of 8th week
  The Constipation Severity Instrument will be used to assess the severity of constipation and associated discomfort. The Constipation Severity Instrument developed by Varma et al. has good internal consistency and test-retest reliability. Kaya et al. found that the Turkish version of The Constipation Severity Instrument has good internal consistency and test-retest reliability. The Constipation Severity Instrument has three subscales: obstructive defecation, colonic inertia, and pain. Higher The Constipation Severity Instrument scores indicate more severe constipation.
The severity of constipation | Change in the severity of constipation from baseline to end of week 8
  The Constipation Scoring System is reliable and valid for the use of constipation severity and consists of 8 domains: frequency of bowel movements, painful emptying attempts, incomplete emptying sensation, abdominal pain, time spent on the toilet per attempt, type of assistance for defecation, number of failed toilet attempts in 24 hours and duration of constipation. Above 15 points is considered constipation.
Gastrointestinal symptom level | Change in gastrointestinal symptom level from baseline to the end of the 8th week
  Gastrointestinal symptom level will be assessed with the "Gastrointestinal Symptom Rating Scale", the reliability and validity of the Turkish version of which was established by Turan et al. This scale is a 7-point Likert-type scale consisting of 15 items. The scale has 5 subscales: abdominal pain, reflux, diarrhea, indigestion and constipation. Higher scores indicate more severe symptoms.
Constipation-related quality of life | Change in constipation-related quality of life from baseline to the end of the 8th week
  The effect of constipation on quality of life will be evaluated with the Patient Assessment of Constipation Quality of Life Questionnaire developed by Marquis et al. Dedeli et al. demonstrated that the Turkish version of the Patient Assessment of Constipation Quality of Life Questionnaire has good internal consistency and test-retest reliability. The questionnaire includes 4 sub-titles: worries and concerns, physical discomfort, psychosocial discomfort and satisfaction.The total score varies between a minimum of 28 and a maximum of 140, and higher scores of Patient Assessment of Constipation Quality of Life Questionnaire indicate more negative effects of constipation on the quality of life.
Patient perception of global change | Patient perception of global change from baseline to the end of 8th week
  The Patient Global Perception of Change Scale, a 7-item scale assessing the perception of change in the impact of constipation and related complaints on the patient's life compared to the start of the study, will be used. The options on this scale are ''much much better'', ''much better'', 'a little better'', ''no change", ''a little worse'', ''much worse'', ''much much worse''.
Abdominal muscle strength | Change in abdominal muscle strength from baseline to the end of the 8th week
  The abdominal muscle strength of the individuals will be assessed by observational/manual muscle strength test. Muscle strength is a widely used anthropometric measurement in the clinic and the measurement standards were developed by Dr. Lovett. Muscle strength is graded on a scale of 0 to 5 by observation or manual resistance.
Functional exercise capacity | Change in functional exercise capacity from baseline to the end of the 8th week
  Functional exercise capacity of the individuals will be evaluated with the 6-minute walk test. The 6-minute walk test (6MWT) is an easy-to-administer, reproducible, data-rich, low-cost and well-tolerated test of walking capacity in which individuals walk at their own pace. During the test, individuals walk for six minutes in an enclosed environment and along a straight corridor of 30 meters in length using standardized commands and encouragement phrases. The distance is recorded in meters. The 6DYT is a test that measures functional exercise capacity, has high construct validity, and is highly correlated with exercise performance and physical activity scales.

CONTACTS AND LOCATIONS:
Overall Officials: Serap ÖZGÜL, Prof, Principal Investigator — Hacettepe University, Department of Physiotherapy and Rehabilitation; Hatice Yasemin BALABAN, Study Director — Hacettepe University, Department of Internal Diseases, Division of Gastroenterology
Locations (2):
- Turkey (Türkiye) (2):
  - Ceren Gursen, Ankara
  - Hacettepe University, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dogan IG, Gursen C, Akbayrak T, Balaban YH, Vahabov C, Uzelpasaci E, Ozgul S. Abdominal Massage in Functional Chronic Constipation: A Randomized Placebo-Controlled Trial. Phys Ther. 2022 Jul 4;102(7):pzac058. doi: 10.1093/ptj/pzac058. PMID 35554601
- [Background] Gao R, Tao Y, Zhou C, Li J, Wang X, Chen L, Li F, Guo L. Exercise therapy in patients with constipation: a systematic review and meta-analysis of randomized controlled trials. Scand J Gastroenterol. 2019 Feb;54(2):169-177. doi: 10.1080/00365521.2019.1568544. Epub 2019 Mar 7. PMID 30843436
- [Background] Sharma A, Rao SSC, Kearns K, Orleck KD, Waldman SA. Review article: diagnosis, management and patient perspectives of the spectrum of constipation disorders. Aliment Pharmacol Ther. 2021 Jun;53(12):1250-1267. doi: 10.1111/apt.16369. Epub 2021 Apr 28. PMID 33909919
- [Background] Pamuk ON, Pamuk GE, Celik AF. Revalidation of description of constipation in terms of recall bias and visual scale analog questionnaire. J Gastroenterol Hepatol. 2003 Dec;18(12):1417-22. doi: 10.1046/j.1440-1746.2003.03155.x. PMID 14675272
- [Background] Lewis SJ, Heaton KW. Stool form scale as a useful guide to intestinal transit time. Scand J Gastroenterol. 1997 Sep;32(9):920-4. doi: 10.3109/00365529709011203. PMID 9299672
- [Background] Varma MG, Wang JY, Berian JR, Patterson TR, McCrea GL, Hart SL. The constipation severity instrument: a validated measure. Dis Colon Rectum. 2008 Feb;51(2):162-72. doi: 10.1007/s10350-007-9140-0. Epub 2008 Jan 3. PMID 18172725
- [Background] McCrea GL, Miaskowski C, Stotts NA, Macera L, Hart SA, Varma MG. Review article: self-report measures to evaluate constipation. Aliment Pharmacol Ther. 2008 Apr;27(8):638-48. doi: 10.1111/j.1365-2036.2008.03626.x. Epub 2008 Jan 23. PMID 18221405
- [Background] Turan N, Ast TA, Kaya N. Reliability and Validity of the Turkish Version of the Gastrointestinal Symptom Rating Scale. Gastroenterol Nurs. 2017 Jan/Feb;40(1):47-55. doi: 10.1097/SGA.0000000000000177. PMID 28134719
- [Background] Marquis P, De La Loge C, Dubois D, McDermott A, Chassany O. Development and validation of the Patient Assessment of Constipation Quality of Life questionnaire. Scand J Gastroenterol. 2005 May;40(5):540-51. doi: 10.1080/00365520510012208. PMID 16036506
- [Background] Bengi G, Yalcin M, Akpinar H, Keskinoglu P, Ellidokuz H. Validity and reliability of the patient assessment of constipation quality of life questionnaire for the Turkish population. Turk J Gastroenterol. 2015 Jul;26(4):309-14. doi: 10.5152/tjg.2015.0185. Epub 2015 Jun 2. PMID 26039000
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Singh SJ, Puhan MA, Andrianopoulos V, Hernandes NA, Mitchell KE, Hill CJ, Lee AL, Camillo CA, Troosters T, Spruit MA, Carlin BW, Wanger J, Pepin V, Saey D, Pitta F, Kaminsky DA, McCormack MC, MacIntyre N, Culver BH, Sciurba FC, Revill SM, Delafosse V, Holland AE. An official systematic review of the European Respiratory Society/American Thoracic Society: measurement properties of field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1447-78. doi: 10.1183/09031936.00150414. Epub 2014 Oct 30. PMID 25359356